CLINICAL TRIAL: NCT04832295
Title: A Study Protocol of the Photo-supported Conversations About Well-being Intervention in People with Stress Related Illness
Brief Title: Photo-supported Conversations About Well-being
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kronoberg County Council (Other Government)
Collaborators: Linnaeus University (Other); Göteborg University (Other); Jonkoping University (Other); Region Jönköping County (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FORSS-847271
Record Dates: First submitted 2021-04-01; First posted 2021-04-05 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Stress Disorder
Keywords: Health promotion
MeSH Terms: conditions — Stress Disorders, Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): Photo-supported conversations about well-being, in addition to care as usual
  Interventions: Other: photo-supported conversations; Other: Care as usual
- Control (Active Comparator): Care as usual
  Interventions: Other: Care as usual

INTERVENTIONS:
Other: photo-supported conversations — Sessions 1-4: Before each of the sessions, the client photographs that which is related to their well-being and send these to the therapist before the session. The therapist enlarges each of the photographs into the size of A4. The conversation departures from the photographs and the client is encouraged to talk about each of them and they ways it relates to their well-being. Potential strategies for everyday life are discussed.
  Session 5-10: short virtual meetings of approximately 15-20 minutes with the aim to follow the client, confirm their process and support them towards increased well-being.
  Session 11: reflecting upon all their previous photographs. Session 12: reflecting future everyday life upon their photographs.
  Other Names: Be Well
  Arms: Intervention
Other: Care as usual — Medication, psychological treatment

SUMMARY:
The aim is to to investigate photo-supported conversations about well-being by the intervention Be WellTM in addition to care as usual within primary care, compared to a control group, for patients with stress-related diagnosis. The intention is to examine the outcomes measures regarding exhaustion, balance of activities in everyday life, client satisfaction, depression and anxiety quality of life, sense of coherence and work ability. The study has been approved by the Regional Ethical Review Board.

The project has a quasi-experimental design using mixed methods. A total of 70 patients (35 to the intervention group and 35 to the control group) will be included. Inclusion criteria are patients with stress-related disorder in primary care, aged 20-67 years, who are on sick leave or risk being on sick leave. Exclusion criteria are severe somatic disorders, neuropsychiatric diagnosis, psychosis and language or cognitive problems that implies difficulties to answer questionnaires.

After informed consent, the intervention group receive, in addition to care as usual, photo-supported conversations about well-being, that is conducted over time for increased training. The intervention involves 12 sessions takes part during 12-15weeks. With cell phones the patients photograph what they relate to well-being in everyday life. The photos are enlarged and used for reflecting conversations with their therapist.

Before and after intervention, and 6 months after intervention the patient meets a project assistant and respond questionnaires as well as qualitative interviews. The control group has the same measure points. Outcome measures are compared with a control group who receive care as usual in primary care. Data will be collected by questionnaires for exhaustion, balance of activities in everyday life, client satisfaction, depression and anxiety, quality of life, sense of coherence and work ability. Qualitative data from interviews about life situation and treatment experiences will also be analyzed. An additional aim is to investigate how therapists experience performing a health promoting intervention, collected from qualitative interviews.

The project is involving the Kronoberg County Council and Jönköping County Council. Gatekeepers will recruit patients and occupational therapists will perform the intervention. The research team comprise of researchers from Kronoberg County Council, Linnaeus University, Jönköping University and University of Gothenburg.

DETAILED DESCRIPTION:
The project has the following research questions:

* How are the participants' work ability, health and well-being affected by the photo-supported intervention?
* Primary outcome is self-rated symptoms of exhaustion.
* Secondary outcomes are self-rated balance of activities in everyday life, client satisfaction, depression and anxiety, quality of life, sense of coherence and work ability.

The interviews deals about:

* How do the participants perceive their life situation, within as well as beyond paid work, before and after the intervention?
* How do the participants perceive their participation photo-supported conversations about well-being intervention (Be Well)?
* How do the therapists perceive the delivery of the intervention "Be Well"?

Non-parametric statistics will be used for analyzing quantitative data. Thematic, phenomenological, qualitative content analyses and semiotic methods will be used for qualitative data.

ELIGIBILITY:
Inclusion Criteria:

* stress related disorder F43.8 (ICD-10)
* stress related disorder F43.9 (ICD-10)
* on sick leave
* risk being on sick leave

Exclusion Criteria:

* severe somatic disorders
* neuropsychiatric diagnosis
* psychosis
* language problems that implies difficulties to answer questionnaires
* cognitive problems that implies difficulties to answer questionnaires

Ages: 20 Years to 67 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2024-10-30 (Actual); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Exhaustion | Up to 9 months after enrollment
  Symptoms of exhaustion measured by Karolinska Exhaustion Disorder Scale (KEDS) (Besèr et al., 2014) min=0 , max=54 , the higher the worse
Work ability | Up to 9 months after enrollment
  Work ability measured by Worker Role Self-assessment (WRS-18) (Ekbladh et al., 2000) min=15 , max= 90, the higher the better

SECONDARY OUTCOMES:
Balance of activities in everyday life | Change from baseline to after treatment, and 6 months
  Balance of activities in everyday life measured by the Occupational Balance questionnaire (OBQ11) (Håkansson et al., 2020) min=0 , max=33, the higher the better
Client Satisfaction | Up to 9 months after enrollment
  Client Satisfaction measured by the Client Satisfaction Questionnaire (CSQ) (Larsen et al., 1979) min=8, max=32, the higher the better
Depression and anxiety | Up to 9 months after enrollment
  Symptoms of Depression and anxiety measured by the Hospital Anxiety and Depression Scale (HADS) (Zigmond & Snaith, 1983), min=0, max=42, the higher the worse
Life quality | Up to 9 months after enrollment
  Quality of life measured with the Manchester Short Assessment of quality of life (MANSA) (Priebe et al., 1999), min=12, max=84, the higher the better
Sense of coherence | Up to 9 months after enrollment
  Sense of coherence measured with the Sense of Coherence Scale (SoC) ((Antonovsky, 1987), min=13, max=91, the higher the better

OTHER OUTCOMES:
Interview | Up to 9 months after enrollment
  situation in everyday life, and what causes stress at home and at work, and what contributes to well-being despite living with stress

CONTACTS AND LOCATIONS:
Overall Officials: Birgitta A Gunnarsson, PhD, Study Chair — Kronoberg County Council
Locations (1):
- Kronoberg County Council, Vaxjo, Sweden

REFERENCES:
- [Derived] Gunnarsson AB, Wagman P, Sternudd HT, Holmberg S, Holmgren K, Horberg U. A study protocol of the photo-supported conversations about the well-being intervention (Be Well) for people with stress related disorders. BMC Psychol. 2021 Aug 21;9(1):123. doi: 10.1186/s40359-021-00625-3. PMID 34419148